CLINICAL TRIAL: NCT01541566
Title: Blood Pressure Control and Compliance to Treatment in Hypertensive Patients With Metabolic Syndrome: a Study Based on Home Blood Pressure Telemonitoring
Brief Title: Blood Pressure Control and Compliance to Treatment in Hypertensive Patients With Metabolic Syndrome: a Study Based on Home Blood Pressure Telemonitoring and Assessment of Psychological Determinants
Acronym: TELEBPMET
Status: Completed | Type: Observational
Sponsor: Italian Institute of Telemedicine (Other)
Collaborators: Bracco Corporate (Industry); Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: TELEBPMET
Record Dates: First submitted 2012-02-17; First posted 2012-03-01 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Arterial Hypertension; Metabolic Syndrome
Keywords: arterial hypertension; metabolic syndrome; home blood pressure; ambulatory blood pressure; office blood pressure; telemedicine
MeSH Terms: conditions — Hypertension; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Home blood pressure telemonitoring: Patients regularly monitoring their blood pressure at home with an electronic validated upper arm device, transmitting blood pressure values at monthly intervals to the doctors office through the Internet.
- Conventional blood pressure measurement: Blood pressure measured only in the doctor's office during quarterly visits, without regular home blood pressure monitoring.

SUMMARY:
The purpose of this study is to assess whether, in patients at high cardiovascular risk (hypertension with metabolic syndrome), long-term (1-year) blood pressure control is most effective when based on home blood pressure telemonitoring and on the feedback to the patient by the doctor between visits, or when based only on blood pressure determination during quarterly office visits.

ELIGIBILITY:
Inclusion Criteria:

* Treated or untreated uncontrolled essential arterial hypertension (office systolic blood pressure >140 or diastolic >90 mmHg + day-time systolic blood pressure >135 or day-time diastolic blood pressure >85 mmHg)
* Metabolic syndrome (ATP III criteria)

Exclusion Criteria:

* Secondary arterial hypertension
* Severe liver or kidney disease
* Immunological disease
* Cardiac arrhythmias

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referring to 12 Hypertension Centers (Hospitals) and suffering from arterial hypertension associated to metabolic syndrome
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with average day-time ambulatory blood pressure <135/85 mmHg | 6 months
Percentage of subjects with average day-time ambulatory blood pressure <135/85 mmHg | 12 months

SECONDARY OUTCOMES:
Psychological determinats of therapeutic adherence | 6 months
Percentage of subjects with office blood pressure <140/90 mmHg | 6 months
Changes in home blood pressure | 6 months
Number of additional medical visits | 6 months
Direct costs of intervention | 6 months
Number of antihypertensive drugs | 6 months
Level of cardiovascular risk by ESC Heart Score and Framingham | 6 months
Target organ damage and outcomes | 6 months
Percentage of patients with metabolic syndrome | 6 months
Psychological determinats of therapeutic adherence | 12 months
Percentage of subjects with office blood pressure <140/90 mmHg | 12 months
Changes in home blood pressure | 12 months
Number of additional medical visits | 12 months
Direct costs of intervention | 12 months
Number of antihypertensive drugs | 12 months
Level of cardiovascular risk by ESC Heart Score and Framingham | 12 months
Target organ damage and outcomes | 12 months
Percentage of patients with metabolic syndrome | 12 months
Percentage of subjects with home blood pressure <135/85 mmHg | 6 months
Percentage of subjects with home blood pressure <135/85 mmHg | 12 months
Changes in 24h blood pressure | 6 months
Changes in 24h blood pressure | 12 months
Changes in office blood pressure | 6 months
Changes in office blood pressure | 12 months
Adherence to treatment | 6 months
Adherence to treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Parati, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (12):
- Italy (12):
  - Policlinico Universitario, Bari, Bari
  - Spedali Civili, Brescia, Brescia
  - Fondazione Maugeri, Lumezzane, Brescia
  - Ospedale San Felice a Cancello, San Felice A Cancello, Caserta
  - Istituto Auxologico Italiano, Milan, Milano
  - Policlinico Universitario, Padua, Padova
  - Ospedale di Broni, Broni, Pavia
  - Fondazione Maugeri, Pavia, Pavia
  - Ospedale Santa Chiara, Pisa, Pisa
  - Ospedale Fatebenefratelli, Roma, Roma
  - Casa di Cura Tortorella, Salerno, Salerno
  - Ospedale di Circolo, Varese, Varese

REFERENCES:
- [Derived] Brugnera A, Compare A, Omboni S, Greco A, Carrara S, Tasca GA, Poletti B, Parati G. Psychological covariates of blood pressure among patients with hypertension and metabolic syndrome. Health Psychol. 2022 Dec;41(12):946-954. doi: 10.1037/hea0001205. Epub 2022 Jul 21. PMID 35862126
- [Derived] Parati G, Omboni S, Compare A, Grossi E, Callus E, Venco A, Destro M, Villa G, Palatini P, Rosei EA, Scalvini S, Taddei S, Manfellotto D, Favale S, De Matteis C, Guglielmi M; TELEBPMET Study Group; Lonati L, Della Rosa F, Tosazzi E, Grandi AM, Maresca AM, Mongiardi C, Mare M, Ricci AR, Cagnoni F, Georgatos J, Besostri V, Ferrari V, Omodeo O, Dorigatti F, Bonso E, Guarnieri C, Muiesan L, Paini A, Stassaldi D, Cinelli A, Bernocchi P, Rocchi S, Magagna A, Ghiadoni L, Del Frate I, Boresi F, Guidi A, Re MA, Pellicciotti L, Florio A, Morani G, Di Lillo S, Ambrosio A, Casciello A, Quaglia M, Forleo C, Ardito MA, Gerunda S, Panunzio M. Blood pressure control and treatment adherence in hypertensive patients with metabolic syndrome: protocol of a randomized controlled study based on home blood pressure telemonitoring vs. conventional management and assessment of psychological determinants of adherence (TELEBPMET Study). Trials. 2013 Jan 23;14:22. doi: 10.1186/1745-6215-14-22. PMID 23343138